CLINICAL TRIAL: NCT00543504
Title: A Phase 1 Study of Bevacizumab in Combination With 1) Sunitinib, 2) Sorafenib, 3) Erlotinib and Cetuximab, 4) Trastuzumab and Lapatinib
Brief Title: Bevacizumab in Multiple Phase I Combinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0638; NCI-2012-01552 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Bevacizumab; Avastin; Sorafenib; BAY 43-9006; Erlotinib; OSI-774; Tarceva; Trastuzumab; Herceptin; Sunitinib; SU011248; Sutent; Cetuximab; Lapatinib; Tykerb; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Erlotinib hydrochloride; GW572016; Sunitinib Malate
MeSH Terms: interventions — Bevacizumab; Sorafenib; Erlotinib Hydrochloride; Trastuzumab; Lapatinib; Sunitinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Bevacizumab + Sunitinib (Experimental): Arm 1: Bevacizumab starting dose 2.5 mg/kg intravenous (IV) over 90 minutes + Sunitinib 12.5 mg orally daily for 4 weeks, then 2 weeks off.
  Interventions: Drug: Bevacizumab; Drug: Sunitinib
- Bevacizumab + Sorafenib (Experimental): Arm 2: Bevacizumab starting dose 2.5 mg/kg intravenous (IV) over 90 minutes + Sorafenib 200 mg by mouth daily for 28 Days
  Interventions: Drug: Bevacizumab; Drug: Sorafenib
- Bevacizumab + Erlotinib + Cetuximab (Experimental): Arm 3: Bevacizumab starting dose 2.5 mg/kg intravenous (IV) over 90 minutes + Erlotinib 50 mg By Mouth Daily for 28 Days + Cetuximab loading dose 100 mg/m² IV and maintenance 75 mg/m² on Days 1, 8, 15, 22.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Cetuximab
- Bevacizumab + Trastuzumab + Lapatinib (Experimental): Arm 4: Bevacizumab starting dose 2.5 mg/kg intravenous (IV) over 90 minutes + Trastuzumab loading dose 2 mg/kg IV then maintenance dose 1 mg/kg IV on Day 1 + Lapatinib 250 mg By Mouth Daily for 21 Days.
  Interventions: Drug: Bevacizumab; Drug: Trastuzumab; Drug: Lapatinib

INTERVENTIONS:
Drug: Bevacizumab — 2.5 mg/kg By Vein Over 90 Minutes.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Sorafenib — 200 mg By Mouth Daily for 28 Days
  Other Names: BAY 43-9006
  Arms: Bevacizumab + Sorafenib
Drug: Erlotinib — 50 mg By Mouth Daily for 28 Days.
  Other Names: Erlotinib hydrochloride; OSI-774; Tarceva
  Arms: Bevacizumab + Erlotinib + Cetuximab
Drug: Trastuzumab — Loading 2 mg/kg by vein then Maintenance 1 mg/kg by vein on Day 1
  Other Names: Herceptin
  Arms: Bevacizumab + Trastuzumab + Lapatinib
Drug: Lapatinib — 250 mg By Mouth Daily for 21 Days.
  Other Names: GW572016; Tykerb
  Arms: Bevacizumab + Trastuzumab + Lapatinib
Drug: Sunitinib — 12.5 mg orally daily for 4 weeks, then 2 weeks off.
  Other Names: Sunitinib Malate; SU011248; Sutent
  Arms: Bevacizumab + Sunitinib
Drug: Cetuximab — Loading 100 mg/m² by vein and Maintenance 75 mg/m² by vein on Days 1, 8, 15, 22
  Arms: Bevacizumab + Erlotinib + Cetuximab

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Avastin™ that can be given in combination with 4 other study drug/drug combinations. It will be given with sunitinib, with sorafenib, with a combination of erlotinib and cetuximab, and with a combination of trastuzumab and lapatinib. The safety and effectiveness of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab (Avastin™) is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels

Sunitinib malate (SutentTM) is designed to block pathways that control important events such as the growth of blood vessels that are vital for the growth of cancer.

Sorafenib (NexavarTM) is designed to block the function of important proteins in cancer cells. These proteins, when active, are in part responsible for the abnormal growth and behavior of cancer cells.

Erlotinib hydrochloride (TarcevaTM) is designed to block the activity of a protein found on the surface of many tumor cells that may control tumor growth and survival. This may stop tumors from growing.

Cetuximab (ErbituxTM) is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the epidermal growth factor receptor (EGFR).

Trastuzumab (HerceptinTM) is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the Her2/neu receptor.

Lapatinib (TykerbTM) is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the Her2/neu receptor and EGFR.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, your doctor will decide which study drugs you will receive based on the disease type and on the drugs you have taken in the past.

Once it is decided which drugs you will receive, you will be enrolled into a group of about 3-6 participants that are receiving the same drug combination. The first group of participants will receive the lowest dose of the drug combination. The next group of participants will receive the next highest dose of the drug combination. The third group will receive an even higher dose than that. This process will continue until the study doctor finds the highest safe dose of the drug combination. The dose that you receive will depend on when you are enrolled in this study and the safety data that is available at that time. The dose that you receive may be lowered if you do not tolerate the study drug combination well.

Once the highest tolerated dose is found for each group, up to 10 more participants will be added to each group at that dose level.

The dose levels testing the study drug combination of bevacizumab with either sunitinib or sorafenib are now closed.

Study Drug Administration:

Avastin™ is given through a needle in your vein. The first infusion is over 90 minutes. The next infusion may be over 60 minutes if the first infusion was well tolerated. If you tolerate the second infusion well, the third infusion may be over 30 minutes. If you take trastuzumab and lapatinib with Avastin™, you will receive Avastin™ every 21 days. If you take cetuximab and erlotinib with Avastin™, you will receive Avastin™ every 14 days.

If you are assigned to take cetuximab and erlotinib, cetuximab will be given by vein once every week. The first time you receive cetuximab, it will be given over 2 hours. All other infusions will be given over 60 minutes. Erlotinib is taken by mouth every day during the 28-day study cycle. You should take erlotinib on an empty stomach either 1 hour before eating or 2 hours after eating.

If you are assigned to take trastuzumab and lapatinib, trastuzumab will be given by vein once every 21-day study cycle. The first infusion will be over 90 minutes. If you handle the infusion well, each additional infusion will be over 30 minutes Lapatinib will be taken by mouth every day for 21 days. You should take lapatinib on an empty stomach either 1 hour before eating or 2 hours after eating.

Study Visits:

Avastin, cetuximab, and erlotinib:

During Cycle 1, you will have a study visit during Weeks 1 and 2. During Cycles 2 and beyond, you will have a study visit during Week 1. At these visits, you will have a physical exam, and blood (about 1 tablespoon) will be drawn for routine tests. If the routine urine test done at screening had abnormal results, urine may be collected for additional routine tests during the study. After 2 cycles, you will have the physical exam every 1-2 months.

Every week, you will have blood drawn (about 2 teaspoons) for routine tests.

During Week 1 of all cycles, you will have urine collected for routine tests.

After every 2 cycles, you will have a CT or MRI scan to check the status of the disease. After 6 months (6 cycles) of study drug treatment, you will have the CT or MRI scan every 2-4 cycles.

Avastin, trastuzumab, and lapatinib:

During Cycle 1, you will have a study visit during Weeks 1 and 2. During Cycles 2 and beyond, you will have a study visit during Week 1. At these visits, you will have a physical exam, and blood (about 1 tablespoon) will be drawn for routine tests. If the routine urine test done at screening had abnormal results, urine may be collected for additional routine tests during the study. After 2 cycles, you will have the physical exam every 1-2 months.

During Week 1 of all cycles, you will have urine collected for routine tests.

After every 2 cycles, you will have a CT or MRI scan to check the status of the disease. After 6 months (8 cycles) of study drug treatment, you will have the CT or MRI scan every 2-4 cycles.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Avastin™, erlotinib, cetuximab, trastuzumab, and lapatinib are all FDA approved and commercially available. Avastin™ is FDA approved for the treatment of colorectal cancer and lung cancer. Erlotinib is FDA approved for the treatment of lung cancer and pancreatic cancer. Cetuximab is FDA approved for the treatment of colorectal cancer and cancer of the head and neck. Trastuzumab is FDA approved for the treatment of breast cancer. Lapatinib is FDA approved for the treatment of breast cancer. The use of these drugs together is investigational and authorized for use in research only.

Up to 354 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or have no standard therapy that induces a CR rate of at least 10% or improves survival by at least three months.
2. Patients must be three weeks from prior cytotoxic therapy; if they have recovered their blood counts to eligibility levels sooner and have no mucositis or other acute toxicities, they may be treated earlier but no sooner than two weeks after their last chemotherapy. Patients must be two weeks or five half lives from biologic therapy, whichever is shorter.
3. ECOG performance status </= 2 (Karnofsky >/= 60%).
4. Patients must have normal organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/=75,000/mL; creatinine </= 3 X ULN; total bilirubin </= 2.0; ALT(SGPT) </= 3 X ULN; Exception for patients with liver metastasis: total bilirubin </= 3 x ULN; ALT(SGPT) </= 5 X ULN. Exception for the bevacizumab + erlotinib + cetuximab arm and the bevacizumab + trastuzumab + lapatinib arm: no minimum absolute neutrophil count or platelet count.
5. The effects of bevacizumab on the developing human fetus are unknown. Angiogenesis is of critical importance to fetal development, and bevacizumab is likely to have adverse consequences in terms of fetal development. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Life expectancy of at least 3 months.
8. Patients with a prior DVT/PE are eligible for treatment if they are receiving or have finished receiving appropriate anticoagulation therapy.

Exclusion Criteria:

1. Patients with hemoptysis within 28 days prior to entering the study.
2. Patients with clinically significant unexplained bleeding within 28 days prior to entering the study.
3. Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg on medication).
4. Patients with clinically significant cardiovascular disease: history of CVA within 6 months, myocardial infarction or unstable angina within 6 months, or unstable angina pectoris.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on Day 1.
6. Pregnant or lactating women.
7. History of hypersensitivity to bevacizumab, murine products, or any component of the formulation.
8. (For patients on the sunitinib treatment arm and the trastuzumab/lapatinib treatment arm only) Left ventricular ejection fraction of less than 50% unless the patient is receiving an angiotensin-converting enzyme (ACE) inhibitor / angiotensin receptor blocker (ARB) and a beta-blocker.
9. (For sorafenib treatment arm only) Hypersensitivity to sorafenib or any component of the formulation.
10. (For erlotinib and cetuximab treatment arm only) History of hypersensitivity to erlotinib or any component of the formulation.
11. (For erlotinib and cetuximab treatment arm only) History of hypersensitivity to cetuximab, murine products, or any component of the formulation.
12. (For trastuzumab and lapatinib treatment arm only) History of hypersensitivity to trastuzumab, Chinese hamster ovary cell proteins, or any component of the formulation.
13. (For trastuzumab and lapatinib treatment arm only) History of hypersensitivity to lapatinib or any component of the formulation.
14. Patients with clinically significant gastrointestinal bleeding within 28 days prior to entering the study.
15. Patients with hemorrhagic brain metastases.
16. Patients with prior abdominal surgery within 30 days prior to entering the study.
17. (For patients on the sunitinib treatment arm and the trastuzumab/lapatinib treatment arm only) Left ventricular ejection fraction of less than 50%, unless the patient is receiving an angiotensin-converting enzyme (ACE) inhibitor / angiotensin receptor blocker (ARB) and a beta-blocker.
18. (For patients on the sunitinib treatment arm and the trastuzumab/lapatinib treatment arm only) QTc prolongation, defined as greater than 440 milliseconds for males, and greater than 460 milliseconds for females.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-10-10 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerable Dose (MTD) of Avastin in combination with 4 other study drug/drug combinations | 28 days
  MTD defined by Dose Limiting Toxicity in first 28 day cycle (induction phase)

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, Dumbrava EI, Jiang Y, Thein KZ, Naing A, Hong DS, Fu S, Piha-Paul SA, Tsimberidou AM, Janku F, Meric-Bernstam F, Kurzrock R, Falchook G. Dual EGFR blockade with cetuximab and erlotinib combined with anti-VEGF antibody bevacizumab in advanced solid tumors: a phase 1 dose escalation triplet combination trial. Exp Hematol Oncol. 2020 Apr 20;9:7. doi: 10.1186/s40164-020-00159-1. eCollection 2020. PMID 32337094
- [Derived] Falchook GS, Moulder SL, Wheler JJ, Jiang Y, Bastida CC, Kurzrock R. Dual HER2 inhibition in combination with anti-VEGF treatment is active in heavily pretreated HER2-positive breast cancer. Ann Oncol. 2013 Dec;24(12):3004-11. doi: 10.1093/annonc/mdt395. Epub 2013 Oct 24. PMID 24158411
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org